**Informed Consent for:** Brief Mindfulness based intervention for Front-Line Medical Staff in the COVID19 Pandemic to improve Psychological Wellbeing, a Randomized Controlled Multicenter Trial.

You are being asked to take part in this study because you are one of our precious front-line medical staff in COVID19 pandemic

Please take your time to make your decision about taking part.

Why is this study being done?

The purpose of this study is to evaluate the effectiveness of brief mindfulness based interventions to frontline HCP wellbeing and in coping for (COVID19).

How many people will take part in the study?

All frontline health care professionals, namely physicians, nurses and respiratory therapist in the 5 largest Eastern province hospitals are invited to participate in the study.

What will happen if I take part in this research study?

You will be invited to answer a pre-intervention questionnaire.

Then will be invited to listen to a 10 minutes audio daily for 2 weeks (you will receive a daily reminder). Then you will be invited to answer a post-intervention questionnaire.

During the study ...

If you choose to take part, you will be "randomized" into one of the study groups described below.

Randomization means that you are put into a group by chance. A computer program will place you in one of the study groups. Neither you nor your study doctor can choose the group you will be in. You will have an equal chance of being placed in either group. Moreover no one will know which group you are assigned to (triple blinded study) except for an electronic file recoreding the allocation.

If you are in group 1 (often called "Arm A"), you will receive brief mindfulness sessions in the audio

If you are in group 2 (often called "Arm B"), you will receive psycho-education sessions in the audio

| Bot | h G | rou | ps |
|-----|-----|-----|--------------|
| DUC | | ıou | $\mathbf{p}$ |

For the duration of this study (2 weeks), you must kindly agree not to share the received audio with anyone

## Study Plan

All data will be anonymously collected to a computer file including the number of times you actually listened to the audio and the duration

How long will I be in the study?

You will be asked to join the study for 2 full weeks

Can I stop being in the study?

Yes. You can decide to stop at any time. Please inform the study team if you are thinking about stopping or decide to stop.

What side effects or risks can I expect from being in the study?

None

Are there benefits to taking part in the study?

Taking part in this study

Might improve your psychological wellbeing

Will my medical information be kept private?

Data are kept in a password-protected database. We will do our best to make sure that the personal information in your medical record will be kept private.

If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

What are the costs of taking part in this study?

There will be no costs to you for participating in this study.

You will not be paid for taking part in this study.

What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study team members may receive your information, but they will not receive your name or other information that would allow them to identify you by name.

Who can answer my questions about the study?

The recruiters

or Dr Amani

Email: qarniamani@icloud.com

I have read it or it has been read to me. I understand the information and have had my questions answered. I agree to take part in this study. By answering the following questions I agree to participate in the study after I had my questions answered.

https://docs.google.com/forms/d/1eNCe9-DDjmlc5GT7o5R37hCTYSeeez6nu8djm-XmR4s/edit